CLINICAL TRIAL: NCT00749866
Title: Can Long Term Nebulised Gentamicin Reduce The Bacterial Burden, Break the Vicious Cycle of Inflammation and Improve Quality of Life in Patients With Bronchiectasis
Brief Title: Long Term Nebulised Gentamicin in Patients With Bronchiectasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Dr Adam Hill; Consultant Physician and Honorary Senior Lecturer, NHS Lothian and University of Edinburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CZB/4/451
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2010-08

CONDITIONS: Bronchiectasis
Keywords: Nebulised antibiotics; Non cystic fibrosis bronchiectasis; Bacterial Load; Inflammation; Quality of Life; Side Effects
MeSH Terms: conditions — Bronchiectasis; Inflammation | interventions — Gentamicins; Sodium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Nebulised Gentamicin
  Interventions: Drug: Gentamicin
- 2 (Placebo Comparator): Nebulised 0.9% Saline
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Gentamicin — Nebulised 80mg twice daily
  Arms: 1
Drug: Saline — Nebulised 4mls 0.9% Saline twice daily
  Arms: 2

SUMMARY:
The hypothesis of this randomized placebo controlled trial is that targeted nebulized gentamicin to the airways will reduce bacterial burden and limit neutrophil airways inflammation. If given long term this will improve symptoms, pulmonary physiology, exercise capacity and health related quality of life with a reduction in exacerbation frequency and health care utilization.

ELIGIBILITY:
Inclusion Criteria:

* Bronchiectasis confirmed by HRCT of the chest
* Clinically stable (not requiring antibiotics for at least 4 weeks preceding the study start date)
* Aged 18-70
* Chronic sputum production > 5 mls for the majority of days in 3 months before enrolment
* Chronically colonized (on at least 2 occasions in the preceding 12 months) whilst clinically stable
* At least two exacerbations in the past year
* Patients able to tolerate a nebulized gentamicin challenge
* FEV1 > 30% predicted
* Smoking < 20 pack year history and ex-smokers >1 year.

Exclusion Criteria:

* Cystic fibrosis
* Emphysema on HRCT chest
* Thoracic surgery within the past 1 year
* Allergic bronchopulmonary aspergillosis
* Poorly controlled asthma ( > 20% diurnal variation in peak expiratory flows despite treatment)
* Unstable angina or uncontrolled congestive cardiac failure
* Active malignancy
* Pregnancy or breast feeding
* Creatinine clearance < 30 mls/minute
* Vestibular instability
* Previous documented intolerance to aminoglycosides

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-05; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Reduction in bacterial load | 1 year

SECONDARY OUTCOMES:
airways and systemic inflammation | 1 year
Spirometry and exercise capacity | 1 year
Exacerbation frequency | 1 year
Health Related Quality of Life | 1 Year
Long term safety with nebulised Gentamicin | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Adam T Hill, MBChB MD, Principal Investigator — NHS Lothian and University of Edinburgh
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, Lothian, United Kingdom

REFERENCES:
- [Derived] Chalmers JD, Smith MP, McHugh BJ, Doherty C, Govan JR, Hill AT. Short- and long-term antibiotic treatment reduces airway and systemic inflammation in non-cystic fibrosis bronchiectasis. Am J Respir Crit Care Med. 2012 Oct 1;186(7):657-65. doi: 10.1164/rccm.201203-0487OC. Epub 2012 Jun 28. PMID 22744718
- [Derived] Murray MP, Govan JR, Doherty CJ, Simpson AJ, Wilkinson TS, Chalmers JD, Greening AP, Haslett C, Hill AT. A randomized controlled trial of nebulized gentamicin in non-cystic fibrosis bronchiectasis. Am J Respir Crit Care Med. 2011 Feb 15;183(4):491-9. doi: 10.1164/rccm.201005-0756OC. Epub 2010 Sep 24. PMID 20870753